CLINICAL TRIAL: NCT05363982
Title: Evaluation of Transcranial Photobiomodulation in Autism Spectrum Disorder: Double-Blind, Placebo-Controlled, Randomized Clinical Study of a Novel Approach
Brief Title: Evaluation of Transcranial Photobiomodulation in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tolga A Ceranoglu, Associate Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021- P- 002646
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Transcranial Photobiomodulation
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial Photobiomodulation (tPBM) Treatment (Active Comparator): Transcranial Photobiomodulation--a noninvasive intervention in which near-infrared light is applied to forebrain.
  Interventions: Device: Transcranial Photobiomodulation (tPBM)
- Placebo/ Sham Treatment (Sham Comparator): The sham treatment will mimic the tPBM procedure, while delivering no light.
  Interventions: Device: Placebo/ Sham

INTERVENTIONS:
Device: Transcranial Photobiomodulation (tPBM) — Transcranial Photobiomodulation (tPBM) is a novel treatment approach based on application of an invisible, non-ionizing electromagnetic wave that results in metabolic modulation in tissues targeted. This intervention consists of exposing bilaterally the frontal brain to the electromagnetic wave that penetrates the skin and skull into brain tissue, is non-invasive and minimally dissipated as thermal energy.
  Other Names:
  Niraxx G1 Headband
  Arms: Transcranial Photobiomodulation (tPBM) Treatment
Device: Placebo/ Sham — The sham treatment will consist of applying all the procedures for the delivery of tPBM, but will not deliver light.
  Arms: Placebo/ Sham Treatment

SUMMARY:
The purpose of this 8-week double-blind randomized placebo-controlled study is to assess the tolerability, safety, and efficacy of tPBM in adult patients with ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by variable presentation of difficulties with socialization, reciprocal communication, and restrictive/repetitive behaviors. An increasingly higher prevalence of ASD is documented in each successive epidemiological survey and the disorder is now estimated to affect up to 2% of youth in the general population. This rise in prevalence is in part attributed to improved recognition of autism in intellectually capable populations.

Currently, there exists no approved treatments for core features of ASD. Instead, available treatment interventions target other psychiatric disorders that frequently co-occur with ASD, including attention, anxiety, and mood disorders.

Transcranial Photobiomodulation (tPBM) is a novel treatment approach based on application of an invisible, non-ionizing electromagnetic wave that results in metabolic modulation in tissues targeted. This intervention consists of exposing bilaterally the frontal brain to the electromagnetic wave that penetrates the skin and skull into brain tissue, is non-invasive and minimally dissipated as thermal energy. The benefits of tPBM are wavelength specific. Electromagnetic wave at 850nm is absorbed by cytochrome c oxidase, a specific chromophore in mitochondria and is associated with increased adenosine triphosphate (ATP) production through the respiratory chain. Ultimately, the increased ATP production leads to increased energy metabolism and activity for the cell, and it is hypothesized that a signaling cascade is also activated promoting cellular plasticity and cytoprotection.

These properties of the tPBM have led to novel therapeutic applications in neurology. In acute ischemic stroke subjects, acute treatment with the tPBM led to significantly better outcome as compared to sham. These results were confirmed in a different cohort of stroke patients with mild to moderate severity of illness. Both studies on stroke subjects showed no significant difference in rate of adverse events, as well as serious adverse events, between the tPBM and sham treated subjects. The tPBM has also been used as a treatment of alopecia and in animal models for methanol-induced retinal toxicity. The tPBM is already widely used for non-invasive assessment of brain function, replacing functional magnetic resonance imaging (fMRI), in studies of infants and young adults, under the name of Near Infrared Spectroscopy) underscoring the relatively low risk of tPBM. The major risk of tPBM when using a laser as the light source is associated with accidental retinal exposure, when beams are projected through the lens, with increased risk of macular degeneration. Light emitting diode (LED) light does not share the same risk level as laser light sources and this clinical trial will have multiple protections to safeguard against this risk.

Proposed treatment with tPBM has been previously studied in patients with Major Depressive Disorder (MDD). MDD has been associated with deficits in brain bioenergetic metabolism. In an experimental model of depression, the mitochondrial respiratory chain was found to be inhibited by chronic stress. Depressed subjects have also significantly lower production of ATP (an energy vector) in their muscle tissue and greater incidence of deletions in their mitochondrial DNA. Data from magnetic resonance spectroscopy in subjects with MDD showed that response to the augmentation of a selective serotonin reuptake inhibitor (SSRI) with triiodothyronine (a thyroid hormone) is associated with restoration of the levels of ATP in the brain. A preliminary open study in 10 depressed subjects has shown that the tPBM was safe, effective and well tolerated. More recently, efficacy and safety of tPBM was also explored in treatment of ASD with promising results and no serious adverse events. In that study, 40 participants received eight 5-min laser light applications to the base of the skull and temporal areas across 4-week period (2 applications per week). A pulsed laser of 635nm was compared to placebo (very weak LEDs) and was shown to be associated with significant improvement in ASD symptoms. Tissue penetration varies at different wavelengths, with 800-850nm range penetrating into deep tissue compared to that of 635nm.

More recently, the investigators completed a prospective, 8-week open-label treatment trial of tPBM in 10 adult patients with moderate to severe level of ASD. Short-term tPBM was well tolerated and was effective in reducing symptom severity of ASD and comorbid ADHD. In addition, tPBM treatment was associated with improvements in executive functions, specifically in functional domains of cognitive flexibility and emotional control, planning and organization, response inhibition and significant improvement in overall function. Treatment with tPBM was well tolerated, and there were no serious adverse events. One subject experienced headache 8 hours after first treatment, and another patient had insomnia after the first treatment episode. Both patients recovered spontaneously and required no changes to study treatments. Current project involves a double-blind randomized clinical trial of tPBM in adult patients with ASD.

The main aim of this 8-week, prospective, placebo (sham) controlled study is to evaluate the efficacy, safety, and tolerability of tPBM with near-infrared light in intellectually capable adults with ASD. Because the tPBM is a non-ionizing radiation, multiple sessions are expected to be safe.

The tPBM treatment can be completed in the comfort of participants' homes, while monitoring their safety and response during scheduled visits. This clinical trial will answer whether tPBM has an effect on ASD symptoms and whether it is safe and acceptable among patients with ASD, for whom frequent visits otherwise would be prohibitive or render it inaccessible.

The advantage of the tPBM treatment approach as compared to pharmacotherapy is that adherence can be easily monitored with device recordings, and the patient is not required to ingest any substance. This proposed study will contribute to answer the question of whether tPBM has an effect on ASD symptoms and whether it is acceptable in minority populations, thus justifying further studies and investments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18 and 59 years of age (inclusive)
* Fulfills Diagnostic and Statistical Manual-5th edition diagnostic criteria for autism spectrum disorder as established by the clinical diagnostic interview.
* Participants with at least moderately severity of ASD symptoms as demonstrated by SRS raw score ≥ 85 and CGI-ASD severity score ≥ 4
* Participants must understand the nature of the study. Participants must be deemed not to have impaired decision-making capacity and must have the capacity to provide direct informed consent. Participants must sign an Institutional Review Board-approved informed consent form before initiation of any study procedures.
* Participants must have a level of understanding sufficient to communicate with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Participant experiencing a major psychiatric disorder will be allowed to participate in the study provided they do not meet any exclusionary criteria.
* Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms with spermicide) if sexually active.
* The subject is willing to participate in this study.

Exclusion Criteria:

* Impaired intellectual capacity (clinically determined). Participants' intellectual capacity will be assessed during the clinical evaluation and determination will be based on intact communicative language, ability to take personal care, history of holding a job and completion of high school (or equivalency credential), and no history of intellectual disability.
* Participant is unable to communicate due to delay in, or total lack of, spoken language development (grossly impaired language skills)
* Clinically unstable psychiatric conditions or judged to be at serious safety risk to self (suicidal risk) or others (within past 30 days).
* Subjects currently (within past 30 days) experiencing significant symptoms of major psychiatric disorders as clinically determined.
* Subjects with an unstable medical condition (that requires clinical attention).
* Active suicidal or homicidal ideation, as determined by clinical screening.
* The subject has a significant skin condition at the procedure sites (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo).
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised arteriovenous malformation, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (verteporfin - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)
* Current treatment with a psychotropic medication on a dose that has not been stable for at least 4 weeks prior to initiating study treatment.
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Atilla Ceranoglu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Achenbach, T. M. and L. A. Rescorla (2003). Manual for ASEBA Adult Forms & Profiles. Burlington, VT, University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Adler LA, Spencer T, Faraone SV, Kessler RC, Howes MJ, Biederman J, Secnik K. Validity of pilot Adult ADHD Self- Report Scale (ASRS) to Rate Adult ADHD symptoms. Ann Clin Psychiatry. 2006 Jul-Sep;18(3):145-8. doi: 10.1080/10401230600801077. PMID 16923651
- [Background] American Psychiatric Association (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA, American Psychiatric Publishing.
- [Background] Ashwood P, Krakowiak P, Hertz-Picciotto I, Hansen R, Pessah I, Van de Water J. Elevated plasma cytokines in autism spectrum disorders provide evidence of immune dysfunction and are associated with impaired behavioral outcome. Brain Behav Immun. 2011 Jan;25(1):40-5. doi: 10.1016/j.bbi.2010.08.003. Epub 2010 Aug 10. PMID 20705131
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators and Centers for Disease Control and Prevention (2012).
- [Background] Blumberg SJ, Bramlett MD, Kogan MD, Schieve LA, Jones JR, Lu MC. Changes in prevalence of parent-reported autism spectrum disorder in school-aged U.S. children: 2007 to 2011-2012. Natl Health Stat Report. 2013 Mar 20;(65):1-11, 1 p following 11. PMID 24988818
- [Background] Cassano P, Cusin C, Mischoulon D, Hamblin MR, De Taboada L, Pisoni A, Chang T, Yeung A, Ionescu DF, Petrie SR, Nierenberg AA, Fava M, Iosifescu DV. Near-Infrared Transcranial Radiation for Major Depressive Disorder: Proof of Concept Study. Psychiatry J. 2015;2015:352979. doi: 10.1155/2015/352979. Epub 2015 Aug 19. PMID 26356811
- [Background] Cassano P, Petrie SR, Hamblin MR, Henderson TA, Iosifescu DV. Review of transcranial photobiomodulation for major depressive disorder: targeting brain metabolism, inflammation, oxidative stress, and neurogenesis. Neurophotonics. 2016 Jul;3(3):031404. doi: 10.1117/1.NPh.3.3.031404. Epub 2016 Mar 4. PMID 26989758
- [Background] Constantino, J. N. and C. P. Gruber (2012). The Social Responsiveness Scale Manual, Second Edition (SRS-2). Los Angeles, CA, Western Psychological Services.
- [Background] Eells JT, Henry MM, Summerfelt P, Wong-Riley MT, Buchmann EV, Kane M, Whelan NT, Whelan HT. Therapeutic photobiomodulation for methanol-induced retinal toxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3439-44. doi: 10.1073/pnas.0534746100. Epub 2003 Mar 7. PMID 12626762
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Endicott, J., R. L. Spitzer, J. L. Fleiss and J. Cohen (1976).
- [Background] Gardner A, Johansson A, Wibom R, Nennesmo I, von Dobeln U, Hagenfeldt L, Hallstrom T. Alterations of mitochondrial function and correlations with personality traits in selected major depressive disorder patients. J Affect Disord. 2003 Sep;76(1-3):55-68. doi: 10.1016/s0165-0327(02)00067-8. PMID 12943934
- [Background] Hamilton, M. (1959).
- [Background] Hamilton, M. (1960).
- [Background] Hollingshead, A. B. (1975). Four Factor Index of Social Status. New Haven, CT, Yale Press.
- [Background] Iosifescu DV, Bolo NR, Nierenberg AA, Jensen JE, Fava M, Renshaw PF. Brain bioenergetics and response to triiodothyronine augmentation in major depressive disorder. Biol Psychiatry. 2008 Jun 15;63(12):1127-34. doi: 10.1016/j.biopsych.2007.11.020. Epub 2008 Jan 22. PMID 18206856
- [Background] Joshi G, Petty C, Wozniak J, Henin A, Fried R, Galdo M, Kotarski M, Walls S, Biederman J. The heavy burden of psychiatric comorbidity in youth with autism spectrum disorders: a large comparative study of a psychiatrically referred population. J Autism Dev Disord. 2010 Nov;40(11):1361-70. doi: 10.1007/s10803-010-0996-9. PMID 20309621
- [Background] Kim EA, Kim BG, Yi CH, Kim IG, Chae CH, Kang SK. Macular degeneration in an arc welder. Ind Health. 2007 Apr;45(2):371-3. doi: 10.2486/indhealth.45.371. PMID 17485886
- [Background] Lampl Y, Zivin JA, Fisher M, Lew R, Welin L, Dahlof B, Borenstein P, Andersson B, Perez J, Caparo C, Ilic S, Oron U. Infrared laser therapy for ischemic stroke: a new treatment strategy: results of the NeuroThera Effectiveness and Safety Trial-1 (NEST-1). Stroke. 2007 Jun;38(6):1843-9. doi: 10.1161/STROKEAHA.106.478230. Epub 2007 Apr 26. PMID 17463313
- [Background] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270
- [Background] Leisman G, Machado C, Machado Y, Chinchilla-Acosta M. Effects of Low-Level Laser Therapy in Autism Spectrum Disorder. Adv Exp Med Biol. 2018;1116:111-130. doi: 10.1007/5584_2018_234. PMID 29956199
- [Background] Mochizuki-Oda N, Kataoka Y, Cui Y, Yamada H, Heya M, Awazu K. Effects of near-infra-red laser irradiation on adenosine triphosphate and adenosine diphosphate contents of rat brain tissue. Neurosci Lett. 2002 May 3;323(3):207-10. doi: 10.1016/s0304-3940(02)00159-3. PMID 11959421
- [Background] National Institute of Mental Health (1985).
- [Background] Rezin GT, Cardoso MR, Goncalves CL, Scaini G, Fraga DB, Riegel RE, Comim CM, Quevedo J, Streck EL. Inhibition of mitochondrial respiratory chain in brain of rats subjected to an experimental model of depression. Neurochem Int. 2008 Dec;53(6-8):395-400. doi: 10.1016/j.neuint.2008.09.012. Epub 2008 Sep 27. PMID 18940214
- [Background] Roth, R. M., P. K. Isquith and G. A. Gioia (2004). Brief-Atm Self report form, Psychological Assessment Resources, Inc.
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Siniscalco D, Schultz S, Brigida AL, Antonucci N. Inflammation and Neuro-Immune Dysregulations in Autism Spectrum Disorders. Pharmaceuticals (Basel). 2018 Jun 4;11(2):56. doi: 10.3390/ph11020056. PMID 29867038
- [Background] Spencer TJ, Adler LA, Meihua Qiao, Saylor KE, Brown TE, Holdnack JA, Schuh KJ, Trzepacz PT, Kelsey DK. Validation of the adult ADHD investigator symptom rating scale (AISRS). J Atten Disord. 2010 Jul;14(1):57-68. doi: 10.1177/1087054709347435. Epub 2009 Sep 30. PMID 19794135
- [Background] StataCorp (2019). Stata Statistical Software: Release 16. College Station, TX.
- [Background] Yamaura M, Yao M, Yaroslavsky I, Cohen R, Smotrich M, Kochevar IE. Low level light effects on inflammatory cytokine production by rheumatoid arthritis synoviocytes. Lasers Surg Med. 2009 Apr;41(4):282-90. doi: 10.1002/lsm.20766. PMID 19347944
- [Background] Zhang Q, Ma H, Nioka S, Chance B. Study of near infrared technology for intracranial hematoma detection. J Biomed Opt. 2000 Apr;5(2):206-13. doi: 10.1117/1.429988. PMID 10938785
- [Background] Zivin, J. A., G. W. Albers, N. Bornstein, T. Chippendale, B. Dahlof, T. Devlin, M. Fisher, W. Hacke, W. Holt, S. Ilic, S. Kasner, R. Lew, M. Nash, J. Perez, M. Rymer, P. Schellinger, D. Schneider, S. Schwab, R. Veltkamp, M. Walker, J. Streeter, E. NeuroThera and I. Safety Trial (2009).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 participants signed consent to participate in the trial, only 30 of those participants were randomized.
Groups:
- Sham: Participants who received sham treatment
- tPBM Treatment: Participants who received tPBM treatment
Period: Overall Study
Arm/Group | Sham | tPBM Treatment
Started | 15 | 15
Completed | 10 | 11
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Population: 15 participants were randomized to the sham treatment, however only 12 were exposed. In the tPBM treatment, 15 participants were randomized to the treatment, however only 13 were exposed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | tPBM Treatment | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian; Native Hawaiian; Pacific Islander | 3 | 0 | 3
  Black/African American | 0 | 1 | 1
  White/Caucasian | 7 | 11 | 18
  Other | 1 | 1 | 2
  Unknown/Not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Adult Behavior Checklist (ABCL) Total T-score
Description: The Adult Behavior Checklist (ABCL) is an observer-rated scale that assesses maladaptive behavioral and emotional problems, social competence and substance use in adults. The item scores are combined into a total score raw score and then transformed into T-scores, ranging from <50 to 80, where a higher T-score indicates a worse outcome. T-scores are calculated with a mean of 50 (population mean) and a standard deviation of 10. This total score reflects overall psychopathology. The outcome reported reflects the change from baseline in ABCL T-scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study medication for at least two weeks. Twenty participants were not included because they either withdrew consent, started a new medication, had the device break and chose not to finish, were not compliant with study procedures, or did not have an informant complete the scale.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 6 | 4
T-score | -4.3 (4.1) | -0.2 (8.3)

2. Secondary Outcome: Change From Baseline in Adult ADHD Investigator Symptom Report Scale (AISRS)
Description: The Adult ADHD Investigator Symptom Report Scale (AISRS) is a clinician-rated scale that assesses ADHD symptoms. It consists of 18 items that are rated on a scale from 0 (not present) to 3 (severe). The item scores are combined into a total score raw score ranging from 0 to 54, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in AISRS scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study medication for at least two weeks. Six participants were not included because they either withdrew consent, started a new medication, had the device break and chose not to finish, were not compliant with study procedures, or were discontinued due to discomfort at treatment site.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 12
score on a scale | -11.8 (8.4) | -8.6 (9.6)

3. Secondary Outcome: Change From Baseline in Adult ADHD Self-Report Scale (ASRS)
Description: The Adult ADHD Self-Report Scale (ASRS) is a patient-rated scale that assesses frequency of ADHD symptoms. It consists of 18 items that are rated on a scale from 0 to 4. The item scores are combined into a total score raw score ranging from 0 to 72, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in ASRS scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study medication for at least two weeks. Five participants were not included because they either withdrew consent, started a new medication, had the device break and chose not to finish, or were not compliant with study procedures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
score on a scale | -13.3 (10.2) | -5.1 (7.4)

4. Secondary Outcome: Change From Baseline in Behavior Rating Inventory of Executive Function-Adult Self Report Version (BRIEF-A) Total T-score
Description: The BRIEF-A is a patient-rated scale that assesses the patient's level of executive function deficits. It consists of 75 items that are rated on a scale from 1 (never) to 3 (often). The item scores are combined into a total score raw score and then transformed into T-scores, ranging from 32 to 91, where a higher T-score indicates a worse outcome. T-scores are calculated with a mean of 50 (population mean) and a standard deviation of 10. This total score is called the Global Executive Composite (GEC) scale and it reflects overall executive functioning. The outcome reported reflects the change from baseline in BRIEF-A Total T-scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
T-score | -13.0 (8.8) | -4.8 (8.9)

5. Secondary Outcome: Improvement in ADHD Symptoms as Assessed by the Clinical Global Impression of Improvement for ADHD (CGI-ADHD-I)
Description: The CGI-ADHD-I is a clinician-rated measure of ADHD symptom improvement since baseline. Improvement scores range from 1 (very much improved) to 7 (very much worse). The outcome reported reflects the number of participants who had CGI-ADHD-I scores of 1 or 2 at study endpoint.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
Patients | 5 | 6

6. Primary Outcome: Participant Improvement in ASD Symptoms as Assessed by the Clinical Global Impression of Improvement for Autism Spectrum Disorder (CGI-ASD-I)
Description: The CGI-ASD-I is a clinician-rated measure of ASD symptom improvement since baseline. Improvement scores range from 1 (very much improved) to 7 (very much worse). The outcome reported reflects the number of participants who had CGI-ASD-I scores of 1 or 2 at study endpoint.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
Participants | 5 | 5

7. Secondary Outcome: Improvement in Anxiety Symptoms as Assessed by the Clinical Global Impression of Improvement for Anxiety (CGI-Anxiety-I)
Description: The CGI-Anxiety-I is a clinician-rated measure of depression symptom improvement since baseline. Improvement scores range from 1 (very much improved) to 7 (very much worse). The outcome reported reflects the number of participants who had CGI-Anxiety-I scores of 1 or 2 at study endpoint.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
Patients | 6 | 8

8. Secondary Outcome: Improvement in Depression Symptoms as Assessed by the Clinical Global Impression of Improvement for Depression (CGI-Depression-I)
Description: The CGI-Depression-I is a clinician-rated measure of depression symptom improvement since baseline. Improvement scores range from 1 (very much improved) to 7 (very much worse). The outcome reported reflects the number of participants who had CGI-Depression-I scores of 1 or 2 at study endpoint.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
Participants | 3 | 6

9. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A)
Description: The Hamilton Anxiety Scale (HAM-A) is a clinician-rated scale that assesses anxiety. It consists of 14 items that are rated on a scale s absent, mild, moderate, severe, or very severe. The item scores are combined into a total score raw score ranging from 17 to 30, where a higher score indicates a worse outcome The outcome reported reflects the change from baseline in HAM-A scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 12
score on a scale | -4.3 (5.4) | -6.0 (5.3)

10. Secondary Outcome: Change From Baseline in Hamilton Depression Scale (HAM-D)
Description: The Hamilton Depression Scale (HAM-D) is a clinician-rated scale that assesses severity of depression in adults. It consists of 21 items that are rated on a scale as absent, mild/trivial, moderate or severe. The item scores are combined into a total score raw score ranging from 0 to 50, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in HAM-D scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 12
score on a scale | -4.3 (4.1) | -5.8 (4.2)

11. Secondary Outcome: Change From Baseline in Massachusetts General Hospital Social Emotional Competence Scale (MGH-SEC)
Description: The MGH-SEC is a clinician-rate scale that assesses change in the frequency and severity of core and associated symptoms of ASD. It consists of 37 items that are rated on a scale from 1 (superior) to 8 (severely). The item scores are combined into a total score which ranges from 37 to 296, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in MGH-SEC scale scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study medication for at least two weeks. Six participants were not included because they either withdrew consent, started a new medication, had the device break and chose not to finish, were not compliant with study procedures, or discontinued the study due to discomfort at the treatment site.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 12
score on a scale | -17.5 (21.4) | -37.6 (26.7)

12. Primary Outcome: Treatment Responders
Description: Treatment responders at study endpoint are defined as those who have a Clinical Global Impression of Improvement for ASD (CGI-ASD-I) score ≤2 and a 25% reduction in score from baseline to study endpoint in the Social Responsiveness Scale-Version 2 (SRS-2) total raw score.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Treatment responders
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
Treatment responders | 2 | 4

13. Primary Outcome: Change From Baseline in Social Responsiveness Scale-2 (SRS-2)
Description: The SRS-2 is a parent-rated scale used to identify the presence and severity of social impairment within the autism spectrum and differentiate it from that which occurs in other disorders. It consists of 65 items that rated on a scale from 1 (not true) to 4 (almost always true). The item scores are recoded by a scorer to 0 (not true) to 3 (almost always true) and combined into a total score which ranges from 0 to 195, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in SRS Total raw scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
score on a scale | -25.3 (20.2) | -25.7 (14.8)

14. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a patient-rated scale that assess evaluate the degree of enjoyment and satisfaction experienced in eight areas of daily functioning. It consists of 16 items that are rated on a scale from 0 (very poor) to 4 (very good). The item scores are combined into a total score raw score ranging from 0 to 64, where a higher score indicates a better quality of life. The outcome reported reflects the change from baseline in Q-LES-Q scores and positive scores represent improvement (i.e., increase in quality of life from baseline).
Time Frame: Baseline to week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham | tPBM Treatment
Number analyzed (Participants) | 12 | 13
score on a scale | 6.4 (9.1) | 3.4 (4.5)

ADVERSE EVENTS:
Time Frame: Baseline to Week 8
Arm/Group | Sham | tPBM Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 10/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham (N=15) | tPBM Treatment (N=15)
Anaphylactic Reaction (General disorders) | 0 | 1 — This event was unexpected and unrelated to study treatment.
Chest pain (exercise induced) (General disorders) | 0 | 1 — This event was unexpected and unrelated to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=15) | tPBM Treatment (N=15)
Headache, migraine, retinal migraine (General disorders) | 2 (2) | 7 (8)
Local/treatment site reactions and device issues: warmth, tingling, pressure, discomfort, wrinkles (General disorders) | 2 (2) | 13 (15)
Sleep problems: disturbed sleep, increased dream recall, insomnia (General disorders) | 4 (4) | 2 (2)
Mood symptoms: flight anxiety, anxiety attack, worsened depression (Psychiatric disorders) | 2 (2) | 1 (1)
Increased forgetfulness, irritability, worsening attention (General disorders) | 1 (1) | 2 (2)
Other: back pain, dizziness, fatigue, Flu, jitteriness, menstrual cramps, allergies (General disorders) | 4 (4) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT05363982/Prot_SAP_000.pdf